CLINICAL TRIAL: NCT01208454
Title: Phase I Study of Vorinostat in Combination With 13-Cis-retinoic Acid in Patients With Refractory/Recurrent Neuroblastoma
Brief Title: Vorinostat and Isotretinoin in Treating Patients With High-Risk Refractory or Recurrent Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02522; NCI-2011-02522 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N2008-02; CDR0000683405; NANT-N2008-02; NANT 08-02; NANT N2008-02 (Other: New Approaches to Neuroblastoma Treatment (NANT)); N2008-02 (Other: CTEP); P01CA081403 (NIH)
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Localized Unresectable Neuroblastoma; Recurrent Neuroblastoma; Regional Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Isotretinoin; Vorinostat

ARMS (1):
- Treatment (isotretinoin and vorinostat) (Experimental): Patients receive isotretinoin PO BID on days 1-14, PO suspension* of vorinostat QD on days 1-4 of course 1, and capsules of vorinostat PO QD on days 1-4 and 8-11 of course 2 and subsequent courses. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  EXPANSION COHORT 1 (=< 21 years of age): Once the MTD has been determined, patients are treated at that dose level as above.
  EXPANSION COHORT 2 (22-30 years of age): Patients receive isotretinoin as above and vorinostat at the MTD on days 1-3 and 8-10.
  Interventions: Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vorinostat

INTERVENTIONS:
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I trial is studying the side effects and the best dose of vorinostat when given together with isotretinoin to see how well it works in treating patients with high-risk refractory or recurrent neuroblastoma. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Isotretinoin may help vorinostat work better by making tumor cells more sensitive to the drug. Giving vorinostat together with isotretinoin may be an effective treatment for neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of vorinostat pediatric suspension administered daily 4 times per week orally for two weeks, in combination with twice daily 13-cis-retinoic acid ([cisRA], isotretinoin) orally for 14 days to children with refractory or recurrent neuroblastoma.

II. To define the toxicities of vorinostat administered in combination with cisRA.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics of vorinostat given as a pediatric suspension.

II. To describe the relationship of vorinostat pharmacokinetics to the occurrence of systemic toxicity.

III. To determine the pharmacokinetics of cisRA given in combination with vorinostat.

IV. To describe histone acetylation levels in peripheral blood mononuclear cells after different doses of vorinostat.

V. To describe, within the context of a Phase I study, the response rate of vorinostat combined with cisRA in patients with recurrent/refractory neuroblastoma.

VI. To describe the toxicity and response rate of vorinostat at the determined maximal tolerated dose combined with cisRA in patients ages 22-30 years of age at study entry with recurrent/refractory neuroblastoma.

OUTLINE: This is a dose-escalation study of vorinostat.

Patients receive isotretinoin orally (PO) twice daily (BID) on days 1-14, PO suspension* of vorinostat once daily (QD) on days 1-4 of course 1, and capsules of vorinostat PO QD on days 1-4 and 8-11 of course 2 and subsequent courses. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

EXPANSION COHORT 1 (=< 21 years of age): Once the maximum-tolerated dose (MTD) has been determined, patients are treated at that dose level as above.

EXPANSION COHORT 2 (22-30 years of age): Patients receive isotretinoin as above and vorinostat at the MTD on days 1-3 and 8-10.

After completion of study therapy, patients are followed up periodically.

NOTE: *Patients less than 10 years of age are encouraged to continue to use oral suspension beyond course 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be =< 21 years of age when registered on study for dose levels -1 to 5 and Expansion Cohort 1; patients age 22-30 years of age at time of study registration are eligible for Expansion Cohort 2
* Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines
* Patients must have high-risk neuroblastoma
* Patients must have at least ONE of the following:

  * Recurrent/progressive disease at any time; biopsy not required, even if partial response to intervening therapy
  * Refractory disease (i.e. less than a partial response to frontline therapy, including a minimum of 4 cycles of chemotherapy); no biopsy is required to document eligibility
  * Persistent disease after at least a partial response to frontline therapy (i.e. patient has had at least a partial response to frontline therapy but still has residual disease by metaiodobenzylguanidine [MIBG] scan, computed tomography [CT]/magentic resonance imaging [MRI], or bone marrow aspirates/biopsies); patients in this category are REQUIRED to have histologic confirmation of viable neuroblastoma from at least one residual site; tumor seen on routine bone marrow morphology is sufficient; bone marrow immunocytology alone is not sufficient for eligibility
* Patients must have at least ONE of the following sites of disease (excluding those patients entered in the Expansion Cohort) :

  * Measurable tumor on MRI or CT scans or X-ray; measurable is defined >= 20 mm in one dimension; for spiral CT defined as >= 10 mm in one dimension; for patients with persistent disease, a biopsy of site seen on CT/MRI must have demonstrated viable neuroblastoma; if the lesion was radiated, then biopsy must be done >= 4 weeks after radiation completed
  * MIBG scan with positive uptake at a minimum of one site; for patients with persistent disease, a biopsy of an MIBG positive site must have demonstrates viable neuroblastoma; if the lesion was radiated, then biopsy must be done >= 4 weeks after radiation completed
  * Bone marrow with tumor cells seen on routine morphology (not by neuron specific enolase [NSE] staining only) of one bone marrow sample of a bilateral aspirate and/or biopsy
* Patients entered in the Expansion Cohorts 1 or 2 who have had a prior relapse are eligible with no measurable or evaluable sites of tumor (i.e. in second complete response)
* Patients must have a life expectancy of at least 6 weeks and a Lansky (=< 16 years) or Karnofsky (> 16 years) score of at least 50
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study enrollment
* Must have received last dose of myelosuppressive chemotherapy at least 3 weeks prior to start of vorinostat; this includes cytotoxic agents given on a low dose metronomic regimen
* Must have received last dose of biologic (anti-neoplastic agent) (includes retinoids) at least 7 days prior to start of vorinostat
* Must have received last dose of monoclonal antibodies at least 7 days or 3 half-lives, whichever is longer, prior to start of vorinostat
* Patients must not have received radiation (small port) for a minimum of two weeks prior to start of vorinostat; for patients with only one site of measurable or evaluable disease, radiation must not have been given to that site unless that site has demonstrated clear progression after radiation
* A minimum of 12 weeks prior to start of vorinostat is required following prior large field radiation therapy (i.e. total body irradiation, craniospinal, whole abdominal, total lung, > 50% marrow space), otherwise a minimum of 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
* Patients are eligible 6 weeks after date of autologous stem cell infusion following myeloablative therapy (timed from start of vorinostat); patients are eligible 6 weeks after date of allogeneic stem cell transplant if without evidence of active graft versus host disease; patients receiving an autologous stem cell infusion to support non-myeloablative therapy are eligible at any time as long as they meet the hematologic and other organ function criteria for eligibility
* A minimum of 6 weeks must have elapsed after 131I-MIBG therapy (timed from start of vorinostat)
* All cytokines or hematopoietic growth factors must be discontinued a minimum of 7 days prior to enrollment on this protocol
* Patients must not be receiving any other anti-cancer agents or radiotherapy at the time of study entry or while on study
* Patients must not be receiving other investigational medications (covered under another investigational new drug [IND]) within 30 days of study entry or while on study
* Since valproic acid has histone deacetylase (HDAC) inhibitory activity, patients must not have received valproic acid within 30 days of study entry
* Prolongation of the corrected QT (QTc) interval has been rarely observed in adults receiving vorinostat; patients must not be receiving azole anti-fungal therapy at the time of study entry or while on protocol therapy; additional agents known to prolong the QTc interval should be avoided unless therapeutic alternative medications are not available
* Patients must not be receiving pentamidine therapy for Pneumocystis pneumonia (PCP) prophylaxis at the time of study entry or while on protocol therapy
* No hematopoietic growth factors within 7 days of enrollment on this protocol
* Patients must not be receiving enzyme-inducing anti-convulsant therapy
* Hemoglobin >= 8 g/dL (transfusion allowed)
* Absolute neutrophil count (ANC) >= 750/uL for patients without marrow metastases at study enrollment; ANC >= 500/uL for patients with marrow metastases at study enrollment
* Platelet count >= 50,000/ul, transfusion independent (no platelet transfusions within 1 week)
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria; patients with marrow disease are not evaluable for hematologic toxicity; if dose limiting hematologic toxicity occurs in two patients, then all subsequent patients enrolled must be evaluable for hematologic toxicity, therefore patients with marrow metastases will be ineligible
* Serum creatinine based on age as follows:

  * 0.8 mg/dL (=< 5 years of age)
  * 1.0 mg/dL (> 5 and =< 10 years of age)
  * 1.2 mg/dL (> 10 and =< 15 years of age)
  * 1.5 mg/dL (> 15 years of age)
* Patient must have a urinalysis with no more than 1+ hematuria and/or no more than 1+ proteinuria
* Total bilirubin =< 1.5 x upper limit of normal for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST}) < 3 x upper limit of normal (note that for ALT, the upper limit of normal for all sites is defined as 45 U/L)
* Alkaline phosphatase =< 2.5 times upper limit of normal
* Normal ejection fraction (>= 55%) documented by either echocardiogram or radionuclide multi gated acquisition scan (MUGA) evaluation OR normal fractional shortening (>= 27%) documented by echocardiogram
* Corrected QT (QTc) interval =< 450 msec
* Serum triglyceride =< 300 mg/dL
* Serum calcium < grade 2
* All post-menarchal females must have a negative beta-human chorionic gonadotropin (HCG); males and females of reproductive age and childbearing potential must use effective contraception for the duration of their participation
* Patients with other ongoing serious medical issues must be approved by the study chair prior to registration
* Patient and/or parent must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnancy, breast feeding, or unwillingness to use effective contraception during the study; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study
* Patients with disease of any major organ system that would compromise their ability to withstand therapy
* Patients with an active or uncontrolled infection; patients on prolonged antifungal therapy are still eligible if they are culture and biopsy negative in suspected radiographic lesions and meet other organ function criteria
* Patients receiving enzyme-inducing anti-convulsants, pentamidine or azole anti-fungal therapy
* Prior treatment with vorinostat combined with cisRA is not allowed; prior therapy with either vorinostat or cis-retinoic acid single agent or combined with alternative agents is allowed
* Patients with a paraben allergy cannot take cisRA preparations containing this compound (i.e., Accutane, Sotret) but are eligible if they can take an alternate preparation without paraben

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity as assessed by NCI CTCAE v. 4.0 | Up to 3 years
  All toxicities observed will be summarized in terms of type (organ affected or laboratory determination), severity (by NCI CTCAE), and attribution. Tables will be created to summarize theses toxicities and side effects by dose level and by course.
MTD of vorinostat, determined according to incidence of dose-limiting toxicities graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | 28 days

SECONDARY OUTCOMES:
Best response, assessed using Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 3 years
Survival | Up to 3 years
Time-to-failure | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie Park, Principal Investigator — New Approaches to Neuroblastoma Treatment (NANT)
Locations (13):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada